CLINICAL TRIAL: NCT04556669
Title: Feasibility and Safety of Anti-PD-L1 Armored Anti-CD22 CAR-T/CAR-TILs Targeting Patients With Solid Tumors
Brief Title: Anti-PD-L1 Armored Anti-CD22 CAR-T/CAR-TILs Targeting Patients With Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Senl_C22P CAR-T/CAR-TIL
Record Dates: First submitted 2020-09-06; First posted 2020-09-21 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Solid Tumor, Adult; Cervical Cancer; Sarcoma; NSCLC
Keywords: CD22; chimeric antigen receptor; solid tumor; tumor infiltration lymphocyte
MeSH Terms: conditions — Uterine Cervical Neoplasms; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD22（aPD-L1）CAR-T cells (Experimental)
  Interventions: Biological: Autologous aPD-L1 armored anti-CD22 CAR T cells

INTERVENTIONS:
Biological: Autologous aPD-L1 armored anti-CD22 CAR T cells — Autologous aPD-L1 armored CD22-targeting CAR T cells

SUMMARY:
This is an open-labeled, single-armed and prospective study, patients with advanced malignant solid tumors will be given with SL22P autologous CAR - T/CAR-TILs cells. The aim of the study is to evaluate the safety and efficacy of SL22P CAR-T cells, including the adverse reaction, pharmacokinetics, and the outcomes of patients.

DETAILED DESCRIPTION:
SL22P is a proprietary product of Senlang Biotechnology. The T cells may be isolated from the peripheral blood or from the tumor tissue. The CAR-T/CAR-TILs cells contains a anti-CD22 CAR structure and also carries a scFv fragment of anti-PD-L1 monoclonal antibody. After autologous SL22P CAR-T/CAR-TILs cells were transplanted back into patients, CAR-T would target CD22+B cells in the blood. This will promote the activation and amplification of CAR+ cells, and secrete anti-PD-L1 scFv outside the cells to regulate the immunity and enhance anti-tumor activity. The CAR-TILs may reduce the severity of the adverse reactions than conventional TILs, which result from the combination of high dose IL-2 infusion.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled, subjects must meet all the following conditions:

1. Volunteer to participate in the clinical study, cooperate with the researcher to carry out the research, and sign the informed consent.
2. 18-75 years old (including boundary value), male or female;
3. Life expectancy ≥ 12 weeks;
4. Patients with ECOG score less than 2
5. All acute toxicity from prior antitumor therapy or surgery is reduced to level 0 to 2.
6. Patients with at least one measurable tumor focus according to recist1.1 standard;
7. Patients with advanced malignant solid tumors who still have disease progression under standard treatment, are intolerant to standard treatments, or lack effective standard treatments, and are pathologically confirmed;
8. Sufficient organ and bone marrow function, defined as follows:

   A) Neutrophil count (ANC) ≥ 1,500/mm3(1.5 × 109/L); B) Platelet count (PLT) ≥ 100,000/mm3 (100 × 109/L); C) Hemoglobin (Hb) ≥ 9 g/dL (90 g/L); D) Serum albumin ≥ 2.8g /dL; E) Serum creatinine ≤ 1.5 times the upper limit of normal value (ULN) or creatinine clearance rate ≥ 50 ml/min; F) Total bilirubin (BIL) ≤ 1.5×ULN, patients with liver metastasis or liver cancer ≤2×ULN; G) AST/SGOT or ALT/SGPT ≤ 2.5×ULN, patients with liver metastasis or liver cancer ≤ 5×ULN; H) International standardized ratio (INR) ≤ 1.5, prothrombin time (PT) and activated partial thrombin time (APTT) ≤ 1.5×ULN.
9. Patients with asymptomatic central nervous system (Central Nervous System, CNS) metastasis, or asymptomatic brain metastases after treatment, must be checked by computed tomography (CT) or magnetic resonance imaging (MRI) without disease progression, stable at least 3 Steroid medication is not required for at least 4 weeks..
10. Male patients and female patients of childbearing age should agree to take effective contraceptive measures from the signing of the informed consent form until 3 months after the last dose.

Exclusion Criteria:

1. Prior therapy with PD-L1 inhibitors
2. Prior therapy as follow:

   A) major surgery within 28 days prior to the first study drug treatment (biopsy required for diagnosis is permitted).

   B) Systemic therapy with immunosuppressive agents within 14 days before the first autologous of study drug, nasal spray and inhaled corticosteroids or physiological doses of steroid hormones are NOT excluded C) Vaccination with live attenuated vaccine within 28 days before the first study drug treatment or planned during the study period and 60 days after the end of the study drug treatment
3. With uncontrollable or symptomatic active central nervous system (CNS) metastasis. Patients with a history of CNS metastasis or spinal cord compression, but if the patient determined to have it stopped by using anticonvulsants and steroids before the first administration and could be clinically stable four weeks later, they may be enrolled in the study.
4. Patients with advanced symptoms, spread to the internal organs, or risk of life-threatening complications in a short-term (including patients with uncontrolled exudate [chest, pericardium, abdominal cavity]).
5. Have any active autoimmune disease or have a history of autoimmune disease and expected recurrence.

   Patients with skin diseases that require no systemic treatment, such as vitiligo, psoriasis, alopecia, type 1 diabetes, or childhood asthma that have been completely alleviated and may be included without any intervention as adults; Asthmatics required medical intervention with bronchodilators are excluded.
6. Had other active malignant tumors within 2 years before entering the study. Skin basal cell that can be treated topically and cured or squamous cell carcinoma, superficial bladder cancer, carcinoma in situ of the cervix, ductal carcinoma in situ of the breast, and papillary thyroid were excluded
7. Patients with seropositive response of Human immunodeficiency virus (HIV) and syphilis, or fail to control the hepatitis B virus or hepatitis C virus infection;
8. Within 6 months before entering the study, the following conditions occurred: myocardial infarction, severe/unstable angina by New York Heart Association Patients with grade 2 or higher cardiac insufficiency and clinically significant supraventricular or ventricular arrhythmia requiring clinical intervention.
9. Severe infection with no effective control.
10. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation is known.
11. Participated in any other drug clinical study within 4 weeks before the first administration, or no more than 5 half-lives before the last study.
12. A history of substance abuse or drug abuse is known.
13. The presence of other serious physical or mental illness or laboratory test abnormalities that may increase the risk of participating in the study or interfere with the results of the study, as well as patients whom the investigator deems inappropriate for participating in the study.

Note: Severe infection refers to sepsis or uncontrolled infection, which can be included in the group only after infection.

Exit criteria :

Withdrawal: This can be divided into investigator performed withdrawal and patient 's voluntary withdrawal from the clinical trial

1. Withdrawal implemented by the investigator: When the patients meets the suspension criteria specified in the protocol during the trial, such as: vital organ dysfunction, drug allergic reaction, poor compliance, worsening of the disease, or serious adverse reactions, it is necessary to stop the trial drug treatment or adopt other treatment methods During treatment, the researcher asked the patients to withdraw from the trial. Due to the differences of patients ' cells, there was a possibility that insufficient number of CAR-T cell can't be prepared.Thus, the investigator judges that the patient needs to withdraw from the study.
2. Patient's withdrawal: such as poor efficacy, intolerance of adverse reactions, hope to adopt other treatment methods, or voluntarily withdraw from the trial without any reason

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
safety evaluation | first three months
  To evaluate the possible adverse reactions recorded within 3 months after SL22P infusion, mainly including the incidence, incidence and severity of skin toxicity, organ toxicity, severe neurotoxicity, cytokine storm and other immunotherapy related toxic reactions (irAEs).

SECONDARY OUTCOMES:
Tmax of cell metabolism | first month
  The highest concentration (Cmax) of anti-CD22 CAR-T cells amplified in peripheral blood; the time to reach the highest concentration (Tmax).
The AUC28d of cell metabolism | first month
  The according area under the curve at 28 days (AUC28d).
PFS evaluation | 12 months
  The researchers evaluated progression-free survival (PFS) according to RECIST V1.1.
OS evaluation | 12 months
  The researchers evaluated overall survival (OS) according to RECIST V1.1.
ORR evaluation | 12 months
  The researchers evaluated objective remission rate (ORR) according to RECIST V1.1.
DoR evaluation | 12 months
  The researchers evaluated remission duration (DoR) according to RECIST V1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyu Wang, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No